CLINICAL TRIAL: NCT04387422
Title: Measurement of Glucose Homeostasis in Human Brain by NMR: Effect of Recurrent Hypoglycemia on Type 1 Diabetes (Aim 2)
Brief Title: Recurrent Hypoglycemia in Type 1 Diabetes (Aim 2)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MED-2019-28365
Record Dates: First submitted 2020-01-31; First posted 2020-05-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 150 mg/dL (Experimental): Hyperglycemia target of 150 mg/dL
  Interventions: Other: Experimental hyperglycemia
- 225 mg/dL (Experimental): Hyperglycemia target of 225 mg/dL
  Interventions: Other: Experimental hyperglycemia
- 300 mg/dL (Experimental): Hyperglycemia target of 300 mg/dL
  Interventions: Other: Experimental hyperglycemia

INTERVENTIONS:
Other: Experimental hyperglycemia — Experimental hyperglycemia with MRI

SUMMARY:
This study will explore the cerebral mechanisms of impaired awareness of hypoglycemia (IAH) in type 1 diabetics following exposure to experimental recurrent hypoglycemia (HG). To induce IAH, patients with T1D identified to have normal awareness of hypoglycemia (NAH) will undergo three 2-hour long hypoglycemic clamps. Neurochemical profiles will be measured by high field MRS before and after induction of IAH. Subject glycemic variability and activity/sleep for 1 week before each study will be monitored as all factors have been shown to alter responses to HG.

DETAILED DESCRIPTION:
The long-term goal of this project is to identify how recurrent hypoglycemia (HG) leads to the clinical syndrome of impaired awareness of hypoglycemia (IAH) in type 1 diabetes (T1D).

This study will test the hypothesis that recurrent HG in T1D leads to an upregulation in brain glucose transport and alterations in glutamatergic and GABAergic tone. The investigators will use MRS methodology that permits evaluation of cerebral cortex and hypothalamus in the same session to simultaneously evaluate the cerebral correlates/mediators of impaired awareness and impaired counterregulatory hormone responses (CRR). High MR data quality and reproducibility will be ensured by using high field MR scanners and technical advances (automated voxel placement, real-time voxel position, frequency, shim updates). Continuous glucose monitoring and actigraphy will be used to chronicle glucose variability and activity/exercise/sleep in the weeks before each experiment to assess the impact of these variables on IAH.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed on clinical or laboratory grounds
* Diabetes duration 2 - 30 years
* Hemoglobin A1C <8.5%

Exclusion Criteria:

* Impaired awareness of hypoglycemia as determined by the Cox and Gold questionnaires
* Pregnant or plan to become pregnant during the study period
* Uncontrolled hypertension (blood pressure > 145/95 mmHg at screening)
* Evidence of autonomic neuropathy (presence of orthostatic hypotension or history of gastroparesis)
* Proliferative retinopathy
* Impaired kidney function (GFR < 45)
* History of myocardial infarction, stroke, seizures, neurosurgical procedures, major depression requiring hospitalization within the last 5 years, arrhythmias
* Current substance abuse
* Use of drugs that can alter glucose metabolism including but not limited to glucocorticoids and niacin, and excluding insulin and glucose lowering drugs used to treat diabetes, as determined by a clinician
* Inability to undergo MRI scanning, including but not limited to unable to remain still in an MRI scanner for more than 30 minutes, claustrophobia, presence of paramagnetic substances or pacemakers in body, weight over 300 lbs
* Unable to complete all study visits or procedures, as determined by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Glucose kinetics during hyperglycemic clamps before and after induction of IAH | 240 Minutes
  A kinetic model of glucose transport through the blood-brain-barrier (BBB) via reversible symmetric Michaelis-Menten kinetics and irreversible utilization in brain tissue will be utilized. The kinetics of glucose transport into and utilization in the frontal cortex will be quantified using dynamic modeling to extract the Michaelis-Menten constants and the maximal rate for glucose transport and utilization. The ratio of maximal transport rate to cerebral metabolic rate of glucose will be estimated for the hypothalamus by steady-state modeling.

SECONDARY OUTCOMES:
Antecedent glycemia concentration | 14 days
  Antecedent glycemia will be evaluated using continuous glucose monitors with particular attention to the percentage of time a participant is above, at, or below target of 80-180 mg/dl and to measures of glycemic variability.
Antecedent physical activity - moderate to vigorous physical activity | 14 days
  Antecedent physical activity and sleep will be evaluated using the data collected by the ActiGraph Link monitors. Activity counts will be set at 15-second epochs and classified into sedentary, light, moderate, and vigorous categories based on Troiano et al. cut points. Participants' average minutes engaged in moderate to vigorous physical activity levels per day will be reported.
Antecedent physical activity - light physical activity | 14 days
  Antecedent physical activity and sleep will be evaluated using the data collected by the ActiGraph Link monitors. Activity counts will be set at 15-second epochs and classified into sedentary, light, moderate, and vigorous categories based on Troiano et al. cut points. Participants' average minutes engaged in light physical activity per day will be reported.
Antecedent physical activity - sedentary time | 14 days
  Antecedent physical activity and sleep will be evaluated using the data collected by the ActiGraph Link monitors. Activity counts will be set at 15-second epochs and classified into sedentary, light, moderate, and vigorous categories based on Troiano et al. cut points. Participants' average minutes engaged in sedentary time per day will be reported.
Antecedent physical activity - energy expenditure | 14 days
  Antecedent physical activity and sleep will be evaluated using the data collected by the ActiGraph Link monitors. Activity counts will be set at 15-second epochs and classified into sedentary, light, moderate, and vigorous categories based on Troiano et al. cut points. Participants' average daily energy expenditure (kilocalories) will be reported.
Antecedent physical activity - sleep quality | 14 days
  Antecedent physical activity and sleep will be evaluated using the data collected by the ActiGraph Link monitors. Activity counts will be set at 15-second epochs and classified into sedentary, light, moderate, and vigorous categories based on Troiano et al. cut points. Participants' average sleep quality will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No